CLINICAL TRIAL: NCT05390099
Title: Evaluation of the Anti-Plaque and Anti-Gingivitis Effects of Moringa Plant Extract and Fluoride Toothpastes Among a Group of Egyptian Children: A Randomized Clinical Trial
Brief Title: Anti-Plaque and Anti-Gingivitis Effects of Moringa Plant Extract and Fluoride Toothpastes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, marwa aly fouad elchaghaby, principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Moringa toothpaste
Record Dates: First submitted 2022-05-20; First posted 2022-05-25 (Actual); Last update posted 2022-05-26 (Actual); Status verified 2022-05

CONDITIONS: Oral Disease
MeSH Terms: conditions — Mouth Diseases

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- moringa plant toothpaste (Experimental)
  Interventions: Drug: Moringa oleifera leaf
- Fluoride toothpaste (Active Comparator)
  Interventions: Drug: Moringa oleifera leaf

INTERVENTIONS:
Drug: Moringa oleifera leaf — Moringa toothpaste

SUMMARY:
The present study aims to assess and compare the anti-plaque and anti-gingivitis effects of Moringa plant extract and Fluoride toothpastes among a group of Egyptian Children.

DETAILED DESCRIPTION:
In the last few years, the use of plant extracts in alternative medicine has evolved widely. Various herbal products, including mouthwash and toothpaste, are now available and have been shown to possess a beneficial effect on oral health .Moringa plant is used to treat various diseases including the treatment of the oral cavity or dentistry .

ELIGIBILITY:
Inclusion Criteria:

* Children of 12-14 years of age.
* Presence of gingivitis-calculus, and plaque (gingival index [GI]score ≥1/plaque index [PI] score ≥1).
* Children willing to participate.
* Children whose parents/caretakers gave informed consent.

Exclusion criteria

* Children having fixed or removable orthodontic appliances or removable prostheses.
* Children suffering from any systemic illness.
* Children who were already using mouthwashes.
* History of oral prophylaxis within 6 months.
* Children using any other oral hygiene aids.

Ages: 12 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2022-04-01 (Actual); Primary Completion 2022-07-01 (Estimated); Study Completion 2022-07-07 (Estimated)

PRIMARY OUTCOMES:
gingival index (Loe and Sillness, 1963) | 6 weeks
  index

SECONDARY OUTCOMES:
plaque index (Sillness and Loe, 1964) | 6 weeks
  index

CONTACTS AND LOCATIONS:
Overall Officials: marwa m elchaghaby, phd, Principal Investigator — marwaaly2003@yahoo.com
Locations (1):
- Cairo university, Giza, Egypt

IPD SHARING:
Plan to Share IPD: No